CLINICAL TRIAL: NCT00969813
Title: A Phase 1, Non-Randomized, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CP-690,550 in Subjects With Hepatic Impairment and Normal Hepatic Function
Brief Title: A Safety and Tolerability Study of CP-690,550 in Subjects With Hepatic Impairment and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: A3921015
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Hepatic Insufficiency
Keywords: Hepatic impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal hepatic function (Experimental)
  Interventions: Drug: CP-690,550
- Mild hepatic impairment (Experimental)
  Interventions: Drug: CP-690,550
- Moderate hepatic impairment (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — Single 10 mg dose of CP-690,550
  Arms: Normal hepatic function
Drug: CP-690,550 — Single 10 mg dose of CP-690,550
  Arms: Mild hepatic impairment
Drug: CP-690,550 — Single 10 mg dose of CP-690,550
  Arms: Moderate hepatic impairment

SUMMARY:
This study is designed to evaluate how CP-690,550 is handled by the body in healthy volunteers who have mild and moderate hepatic impairment compared to healthy volunteers with normal hepatic function. This study will also evaluate the safety and tolerability of CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who have normal liver function, and subjects who have either mild or moderate liver impairment.

Exclusion Criteria:

* Subjects with severe liver impairment
* Subjects who have weakened immune systems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of CP-690,550 in subjects with hepatic impairment compared to subjects with normal hepatic function | 3 days

SECONDARY OUTCOMES:
Safety and tolerability of CP-690,550 in subjects with hepatic impairment compared to subjects with normal hepatic function | 10-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- [Derived] Lawendy N, Lamba M, Chan G, Wang R, Alvey CW, Krishnaswami S. The effect of mild and moderate hepatic impairment on the pharmacokinetics of tofacitinib, an orally active Janus kinase inhibitor. Clin Pharmacol Drug Dev. 2014 Nov;3(6):421-7. doi: 10.1002/cpdd.143. Epub 2014 Oct 1. PMID 27129117
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921015&StudyName=A%20Safety%20and%20Tolerability%20Study%20of%20CP-690%2C550%20in%20Subjects%20with%20Hepatic%20Impairment%20and%20Normal%20Hepatic%20Function